CLINICAL TRIAL: NCT05602311
Title: Effects of General Anesthesia on Brain Functional Connectivity and Cognition in Children With Potential Neurological Damage
Brief Title: Effects of General Anesthesia on Brain FC and Cognition in Children With Potential Neurological Damage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lai Jiang, Chief physician of Department of Anesthesia and Critical Care, Xinhua Hospital affiliated to Shanghai Jiao Tong University, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-22-006
Record Dates: First submitted 2022-08-15; First posted 2022-11-02 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: pediatric anesthesia; POCD; fNIRS; functional connectivity
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Anesthetics, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group SDB: Children were divided into two groups according to whether they had SDB, group SDB: experimental group (SDB children), group control: control group (typical development children)
  Interventions: Drug: General anesthetic
- Group control: Children were divided into two groups according to whether they had SDB, group SDB: experimental group (SDB children), group control: control group (typical development children)
  Interventions: Drug: General anesthetic

INTERVENTIONS:
Drug: General anesthetic — Monitoring the changes of brain functional connectivity and assess cognition in two groups after general anesthesia

SUMMARY:
Postoperative Cognitive Dysfunction(POCD)is a common postoperative complications, existing clinical research focused on the adult patients, ignoring that the developing human brain with underlying neurological impairments may be at higher risk for cognitive impairment, so we need a prospective study, observe this kind of "special groups" in the brain structure and function of before and after general anesthesia, To determine the susceptibility to neurotoxicity of general anesthesia drugs.

DETAILED DESCRIPTION:
Cognitive disorder refers to the abnormal or hindering of people's cognition of learning, memory, thinking, spirit, emotion and psychology, etc. In severe cases, aphasia, agnosia and apraxia will occur. In general, any factors that cause functional and structural abnormalities of the cerebral cortex can lead to cognitive impairment, and surgical anesthesia is one of the factors. Postoperative Cognitive Dysfunction (POCD) broadly refers to the temporary deterioration of cognitive function related to surgery. The diagnosis requires preoperative (as baseline) and postoperative neuropsychological tests, and the degree of postoperative cognitive decline can be determined by comparing the results of preoperative and postoperative tests. Numerous studies have shown that elderly patients are at higher risk for POCD after surgery and anesthesia. Although the neurotoxic effects of narcotic drugs on young neuronal cells have also been extensively discussed in recent years, the current lack of studies on POCD in children is in sharp contrast to the large literature on POCD in adults. The potential impact of general anesthesia on POCD in these younger populations, especially preschool and school age children, is largely unknown due to insufficient clinical evidence.

The effects of general anesthesia on cognitive function in children are complex and controversial. Although a considerable number of animal studies have shown a link between general anesthesia and short-term or long-term neurocognitive impairment in animals, extrapolation of the results to humans remains difficult. Children's central nervous system has not yet mature, general anesthetics on its neurotoxic effect is still not clear, the existing clinical research results differ: some studies have shown that experience a single brief general anesthesia on children and long-term neurological development has no obvious negative impact, some research said general anesthesia to impaired cognitive function in children, especially after the experience again and again, long time exposure to anesthesia. However, few clinical studies have investigated the effects of general anesthesia on cognitive function in children with underlying neurological impairment. Are the effects of general anesthesia drugs on brain function and brain network structure in this "special population" with neurofragility different from those in children without neurological damage risk? Whether general anesthesia can increase the risk of postoperative cognitive impairment or aggravate the existing cognitive dysfunction in this "special population" deserves further study.

Obstructive sleep disordered breathing (SDB) in children is a spectrum of continuous nocturnal breathing disorders characterized by more than airway obstruction and varying degrees of abnormal gas exchange. The mildest of the SDB is Primary Snoring (PS), which is characterized by habitual snoring (often defined as snoring more than three times per week) but few respiratory events (<1 event/hour), decreased oxygen saturation, or slight awakening due to labored breathing; The most severe condition is Obstructive Sleep Apnea (OSA), which is characterized by recurrent episodes of complete or partial airway obstruction, resulting in decreased oxygen saturation at night and or sleep awakenings.

Children with OSA often present with snoring, sleep structure disorder, frequent oxygen desaturation, daytime sleepiness, attention deficit disorder and other symptoms. Adenoid and tonsillar hypertrophy is considered to be the most common cause of SDB in children. A large number of studies have shown that SDB patients have decreased cognitive function and learning ability, including attention, executive function, language learning and memory function. In addition, it has been reported that SDB children have structural changes in different brain regions, especially the hippocampus and frontal cortex, in addition to cognitive impairment. Some scholars believe that SDB may be an independent risk factor for postoperative cognitive impairment.

The human brain can be regarded as a network of interconnected structures and synchronized functions. With the change of the functional state of the brain, the brain network is in dynamic change. The use of neuroimaging techniques (such as functional nuclear magnetic resonance, functional near infrared spectroscopy, etc.) and electrophysiological techniques (such as electroencephalography) can reconstruct the human brain network, which is conducive to the further study of brain structure and function. Based on these techniques, a growing number of researchers have found resting-state or task-state brain network changes in children with neuropsychiatric disorders with different patterns of cognitive and behavioral disorders, such as autism, attention deficit hyperactivity disorder, and epilepsy. In addition to brain network changes occurring in pathological conditions, many drugs that directly act on the central nervous system can also cause brain network changes, and general anesthesia drugs are one of them.

The brain network changes in adults and children under maintenance of general anesthesia, which may be a macroscopic reflection of the molecular mechanism of consciousness loss caused by general anesthesia. Previous studies have shown that the prefrontal and frontal functional connectivity of electroencephalogram in children under maintenance of general anesthesia increases, while the parieto-occipital functional connectivity decreases.

Thus, cognitive impairment is often accompanied by the change of brain network, and general anesthesia on brain networks may also be affected, in view of some adult clinical study shows that preoperative neurocognitie dysfunction or potential risk of cognitive dysfunction in patients with postoperative cognitive function damage probability increases, we hypothesized that: Children with SDB who are still in brain development and have a high risk of neurological injury belong to the "special population" who are more susceptible to the neurotoxicity of general anesthesia drugs. It is hypothesized that the susceptibility to neurotoxicity of general anesthesia drugs in this population is due to the more obvious inhibitory effect of general anesthesia drugs on the existing brain network connectivity. In diseases and general anesthetics on brain network, under the "double whammy" of SDB in children with the normal development of children after general anesthesia operation may face a higher risk of POCD, need to be evaluate cognitive function before and after exposure to general anesthesia, in order to make clear the SDB patients with preoperative cognitive development situation and short-term changes in cognitive function after general anesthesia surgery, At the same time, the changes of brain network before and after anesthesia in children with SDB were observed, and whether the changes of brain network were correlated with the changes of cognitive function was analyzed, so as to try to explain the increased susceptibility to neurotoxicity of general anesthesia in children with neurological injury risk.

Above all，POCD is a common postoperative complications, existing clinical research focused on the adult patients, ignoring that the developing human brain with underlying neurological impairments may be at higher risk for cognitive impairment, so we need a prospective study, observe this kind of "special groups" in the brain structure and function of before and after general anesthesia, To determine the susceptibility to neurotoxicity of general anesthesia drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4 to 10 years old, both sexes;
2. Apgar score ≥8 at birth;
3. ASA (American Society of Anesthesiologists Physical Condition Rating) ⅰ-ⅲ;
4. to be treated with SDB under general anesthesia;
5. His legal guardian has signed the informed consent -

Exclusion Criteria:

1. Age < 4 years old; or age >10 years old;
2. suffering from serious heart, lung and brain diseases;
3. History of dystocia or perinatal cerebral ischemia and hypoxia;
4. Gestational age at birth ≤32 weeks;
5. Confirmed or suspected neurological retardation or hearing and vision abnormalities;
6. suffering from malignant tumor;
7. had received general anesthesia or deep sedation before enrollment

Ages: 4 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Children aged 4-10 years who planned to undergo surgical treatment or examination under general anesthesia in Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine from August 1, 2022 to November 1, 2022 were recruited. Children with SDB who planned to undergo tonsillectomy or adenoidectomy under general anesthesia were selected as the experimental group. According to the age and gender of the children participating in the study, children aged 4-10 years with non-SDB who planned to undergo short surgery under general anesthesia were selected as the control group according to the 1:1 matching principle. Subjects who met the inclusion criteria could enter the study after signing the informed consent form by their legal guardians.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in the scores of Wechsler intelligence scale | The 1 day before surgery；24 hours after surgery
  The scores of Wechsler intelligence scale before operation and 1 day after operation were compared between the two groups.
The incidence of POCD | up to 24 hours after surgery
  The incidence of POCD was calculated by Z-score method

SECONDARY OUTCOMES:
comparison of functional connectivity | up to 5 minutes
  The changes of brain functional connectivity were compared between the two groups under two states of consciousness (awake and anesthesia)
Correlation between fNIRS brain function connectivity and cognitive function changes | one day before surgery and 24 hours after surgery
  The correlation between cognitive function changes and brain functional connectivity, age and anesthesia time were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: lai jiang, Dr., Principal Investigator — Xinhua Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Department of Anesthesia, Shanghai Xinhua hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
No decision on sharing intellectual property rights

REFERENCES:
- [Background] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989
- [Background] Evered LA, Silbert BS. Postoperative Cognitive Dysfunction and Noncardiac Surgery. Anesth Analg. 2018 Aug;127(2):496-505. doi: 10.1213/ANE.0000000000003514. PMID 29889707
- [Background] Zhang D, Ying J, Ma X, Gao Z, Chen H, Zhu S, Shi L, Lu X. Social Cognitive Dysfunction in Elderly Patients After Anesthesia and Surgery. Front Psychol. 2020 Sep 24;11:541161. doi: 10.3389/fpsyg.2020.541161. eCollection 2020. PMID 33071859
- [Background] Ehsani R, Djalali Motlagh S, Zaman B, Sehat Kashani S, Ghodraty MR. Effect of General Versus Spinal Anesthesia on Postoperative Delirium and Early Cognitive Dysfunction in Elderly Patients. Anesth Pain Med. 2020 Aug 8;10(4):e101815. doi: 10.5812/aapm.101815. eCollection 2020 Aug. PMID 33134142
- [Background] Kulason K, Nouchi R, Hoshikawa Y, Noda M, Okada Y, Kawashima R. Indication of Cognitive Change and Associated Risk Factor after Thoracic Surgery in the Elderly: A Pilot Study. Front Aging Neurosci. 2017 Dec 5;9:396. doi: 10.3389/fnagi.2017.00396. eCollection 2017. PMID 29259553
- [Background] Ikonomidou C, Bosch F, Miksa M, Bittigau P, Vockler J, Dikranian K, Tenkova TI, Stefovska V, Turski L, Olney JW. Blockade of NMDA receptors and apoptotic neurodegeneration in the developing brain. Science. 1999 Jan 1;283(5398):70-4. doi: 10.1126/science.283.5398.70. PMID 9872743
- [Background] Ji C, Ni Q, Chen W, Yang Z, Ma D. General anesthetic neurotoxicity in the young: Mechanism and prevention. Neurosci Biobehav Rev. 2019 Dec;107:883-896. doi: 10.1016/j.neubiorev.2019.10.003. Epub 2019 Oct 10. PMID 31606415
- [Background] Amrock LG, Starner ML, Murphy KL, Baxter MG. Long-term effects of single or multiple neonatal sevoflurane exposures on rat hippocampal ultrastructure. Anesthesiology. 2015 Jan;122(1):87-95. doi: 10.1097/ALN.0000000000000477. PMID 25289484
- [Background] Davidson AJ, Disma N, de Graaff JC, Withington DE, Dorris L, Bell G, Stargatt R, Bellinger DC, Schuster T, Arnup SJ, Hardy P, Hunt RW, Takagi MJ, Giribaldi G, Hartmann PL, Salvo I, Morton NS, von Ungern Sternberg BS, Locatelli BG, Wilton N, Lynn A, Thomas JJ, Polaner D, Bagshaw O, Szmuk P, Absalom AR, Frawley G, Berde C, Ormond GD, Marmor J, McCann ME; GAS consortium. Neurodevelopmental outcome at 2 years of age after general anaesthesia and awake-regional anaesthesia in infancy (GAS): an international multicentre, randomised controlled trial. Lancet. 2016 Jan 16;387(10015):239-50. doi: 10.1016/S0140-6736(15)00608-X. Epub 2015 Nov 4. PMID 26507180
- [Background] McCann ME, de Graaff JC, Dorris L, Disma N, Withington D, Bell G, Grobler A, Stargatt R, Hunt RW, Sheppard SJ, Marmor J, Giribaldi G, Bellinger DC, Hartmann PL, Hardy P, Frawley G, Izzo F, von Ungern Sternberg BS, Lynn A, Wilton N, Mueller M, Polaner DM, Absalom AR, Szmuk P, Morton N, Berde C, Soriano S, Davidson AJ; GAS Consortium. Neurodevelopmental outcome at 5 years of age after general anaesthesia or awake-regional anaesthesia in infancy (GAS): an international, multicentre, randomised, controlled equivalence trial. Lancet. 2019 Feb 16;393(10172):664-677. doi: 10.1016/S0140-6736(18)32485-1. Epub 2019 Feb 14. PMID 30782342
- [Background] Sun LS, Li G, Miller TL, Salorio C, Byrne MW, Bellinger DC, Ing C, Park R, Radcliffe J, Hays SR, DiMaggio CJ, Cooper TJ, Rauh V, Maxwell LG, Youn A, McGowan FX. Association Between a Single General Anesthesia Exposure Before Age 36 Months and Neurocognitive Outcomes in Later Childhood. JAMA. 2016 Jun 7;315(21):2312-20. doi: 10.1001/jama.2016.6967. PMID 27272582
- [Background] Warner DO, Zaccariello MJ, Katusic SK, Schroeder DR, Hanson AC, Schulte PJ, Buenvenida SL, Gleich SJ, Wilder RT, Sprung J, Hu D, Voigt RG, Paule MG, Chelonis JJ, Flick RP. Neuropsychological and Behavioral Outcomes after Exposure of Young Children to Procedures Requiring General Anesthesia: The Mayo Anesthesia Safety in Kids (MASK) Study. Anesthesiology. 2018 Jul;129(1):89-105. doi: 10.1097/ALN.0000000000002232. PMID 29672337
- [Background] Zaccariello MJ, Frank RD, Lee M, Kirsch AC, Schroeder DR, Hanson AC, Schulte PJ, Wilder RT, Sprung J, Katusic SK, Flick RP, Warner DO. Patterns of neuropsychological changes after general anaesthesia in young children: secondary analysis of the Mayo Anesthesia Safety in Kids study. Br J Anaesth. 2019 May;122(5):671-681. doi: 10.1016/j.bja.2019.01.022. PMID 30982593
- [Background] Shi Y, Dykhoff HJ, Guevara LRH, Sangaralingham LR, Schroeder DR, Flick RP, Zaccariello MJ, Warner DO. Moderators of the association between attention-deficit/hyperactivity disorder and exposure to anaesthesia and surgery in children. Br J Anaesth. 2021 Nov;127(5):722-728. doi: 10.1016/j.bja.2021.07.025. Epub 2021 Sep 6. PMID 34503832
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Lumeng JC, Chervin RD. Epidemiology of pediatric obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):242-52. doi: 10.1513/pats.200708-135MG. PMID 18250218
- [Background] Katz ES, D'Ambrosio CM. Pathophysiology of pediatric obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):253-62. doi: 10.1513/pats.200707-111MG. PMID 18250219
- [Background] Buratti L, Viticchi G, Baldinelli S, Falsetti L, Luzzi S, Pulcini A, Petrelli C, Provinciali L, Silvestrini M. Sleep Apnea, Cognitive Profile, and Vascular Changes: An Intriguing Relationship. J Alzheimers Dis. 2017;60(3):1195-1203. doi: 10.3233/JAD-170445. PMID 28984599
- [Background] Bourke R, Anderson V, Yang JS, Jackman AR, Killedar A, Nixon GM, Davey MJ, Walker AM, Trinder J, Horne RS. Cognitive and academic functions are impaired in children with all severities of sleep-disordered breathing. Sleep Med. 2011 May;12(5):489-96. doi: 10.1016/j.sleep.2010.11.010. Epub 2011 Apr 13. PMID 21493135
- [Background] Slim M, Westmacott R, Toutounji S, Singh J, Narang I, Weiss S, Krishnan P, Grbac E, Surmava AM, Andres K, MacGregor D, deVeber G, Moharir M, Dlamini N. Obstructive sleep apnea syndrome and neuropsychological function in pediatric stroke. Eur J Paediatr Neurol. 2020 Mar;25:82-89. doi: 10.1016/j.ejpn.2019.11.006. Epub 2019 Nov 21. PMID 31787553
- [Background] Cha J, Zea-Hernandez JA, Sin S, Graw-Panzer K, Shifteh K, Isasi CR, Wagshul ME, Moran EE, Posner J, Zimmerman ME, Arens R. The Effects of Obstructive Sleep Apnea Syndrome on the Dentate Gyrus and Learning and Memory in Children. J Neurosci. 2017 Apr 19;37(16):4280-4288. doi: 10.1523/JNEUROSCI.3583-16.2017. Epub 2017 Mar 20. PMID 28320844
- [Background] Zhao J, Han S, Zhang J, Wang G, Wang H, Xu Z, Tai J, Peng X, Guo Y, Liu H, Tian J, Jin X, Zheng L, Zhang J, Ni X. Association between mild or moderate obstructive sleep apnea-hypopnea syndrome and cognitive dysfunction in children. Sleep Med. 2018 Oct;50:132-136. doi: 10.1016/j.sleep.2018.04.009. Epub 2018 Jun 9. PMID 30036785
- [Background] Daurat A, Sarhane M, Tiberge M. [Obstructive sleep apnea syndrome and cognition: A review]. Neurophysiol Clin. 2016 Jun;46(3):201-15. doi: 10.1016/j.neucli.2016.04.002. Epub 2016 Jun 16. French. PMID 27321089
- [Background] Strutz P, Tzeng W, Arrington B, Kronzer V, McKinnon S, Ben Abdallah A, Haroutounian S, Avidan MS. Obstructive sleep apnea as an independent predictor of postoperative delirium and pain: protocol for an observational study of a surgical cohort. F1000Res. 2018 Mar 15;7:328. doi: 10.12688/f1000research.14061.2. eCollection 2018. PMID 30026927
- [Background] Uddin LQ, Dajani DR, Voorhies W, Bednarz H, Kana RK. Progress and roadblocks in the search for brain-based biomarkers of autism and attention-deficit/hyperactivity disorder. Transl Psychiatry. 2017 Aug 22;7(8):e1218. doi: 10.1038/tp.2017.164. PMID 28892073
- [Background] Guo X, Duan X, Chen H, He C, Xiao J, Han S, Fan YS, Guo J, Chen H. Altered inter- and intrahemispheric functional connectivity dynamics in autistic children. Hum Brain Mapp. 2020 Feb 1;41(2):419-428. doi: 10.1002/hbm.24812. Epub 2019 Oct 10. PMID 31600014
- [Background] Lin H, Lin Q, Li H, Wang M, Chen H, Liang Y, Bu X, Wang W, Yi Y, Zhao Y, Zhang X, Xie Y, Du S, Yang C, Huang X. Functional Connectivity of Attention-Related Networks in Drug-Naive Children With ADHD. J Atten Disord. 2021 Feb;25(3):377-388. doi: 10.1177/1087054718802017. Epub 2018 Sep 27. PMID 30259777
- [Background] Li R, Wang L, Chen H, Guo X, Liao W, Tang YL, Chen H. Abnormal dynamics of functional connectivity density in children with benign epilepsy with centrotemporal spikes. Brain Imaging Behav. 2019 Aug;13(4):985-994. doi: 10.1007/s11682-018-9914-0. PMID 29956102
- [Background] Puglia MP, Vlisides PE, Kaplan CM, Jewell ES, Therrian M, Mashour GA, Li D. Constrained Functional Connectivity Dynamics in Pediatric Surgical Patients Undergoing General Anesthesia. Anesthesiology. 2022 Jul 1;137(1):28-40. doi: 10.1097/ALN.0000000000004221. PMID 35363264
- [Background] Kline RP, Pirraglia E, Cheng H, De Santi S, Li Y, Haile M, de Leon MJ, Bekker A; Alzheimer's Disease Neuroimaging Initiative. Surgery and brain atrophy in cognitively normal elderly subjects and subjects diagnosed with mild cognitive impairment. Anesthesiology. 2012 Mar;116(3):603-12. doi: 10.1097/ALN.0b013e318246ec0b. PMID 22293721
- [Background] Tasbihgou SR, Absalom AR. Postoperative neurocognitive disorders. Korean J Anesthesiol. 2021 Feb;74(1):15-22. doi: 10.4097/kja.20294. Epub 2020 Jul 6. PMID 32623846
- [Background] Evered L, Scott DA, Silbert B, Maruff P. Postoperative cognitive dysfunction is independent of type of surgery and anesthetic. Anesth Analg. 2011 May;112(5):1179-85. doi: 10.1213/ANE.0b013e318215217e. Epub 2011 Apr 7. PMID 21474666